CLINICAL TRIAL: NCT00102336
Title: A Randomized, Placebo Controlled Study Evaluating the Efficacy and Safety of AMG 531 Treatment of Thrombocytopenic Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP) Prior to Splenectomy
Brief Title: AMG 531 Treatment of Thrombocytopenic Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP) Prior to Splenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030212
Record Dates: First submitted 2005-01-27; First posted 2005-01-28 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Thrombocytopenia; Idiopathic Thrombocytopenic Purpura
Keywords: immune (idiopathic) thrombocytopenic purpura; pre-splenectomy; ITP; Thrombopenia
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AMG 531 (Experimental): Active investigational product
  Interventions: Biological: AMG 531
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AMG 531 — Weekly subcutaneous dosing based on screening weight and platelet count. Starting dose is at 1mcg/kg up to a maximum dose of 15mcg/kg. AMG 531 is supplied in a 5 mL single use glass vial as a sterile, white, preservative-free, lyophilized powder.
  Arms: AMG 531
Drug: Placebo — Weekly subcutaneous dosing based on screening weight and platelet count. Starting dose is at 1mcg/kg up to a maximum dose of 15mcg/kg. Placebo is supplied as a lyophilized power in a 5 mL single use glass vial.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of AMG 531 in the treatment of thrombocytopenia in subjects with ITP as measured by the platelet response. This study will also evaluate changes in Patient Reported Outcomes and Health Resource Utilization due to treatment with AMG 531.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ITP according to American Society of Hematology (ASH) guidelines (Appendix F)
* Have completed as least 1 prior treatment for ITP (e.g., prednisone)
* Subjects greater than 60 years of age must have a documented history of chronic ITP with a bone marrow report to confirm the diagnosis
* The platelet count (calculated from the mean of the 2 counts taken during the screening and pre-treatment periods) must be:

  *less than 30 x 10^9/L for those subjects not receiving any ITP therapy, with no count greater than 35 x 10^9/L *less than 50 x 10^9/L for those subjects receiving a constant dose schedule of corticosteroids, azathioprine or danazol with no count greater than 55 x 10^9/L
* A serum creatinine concentration less than or equal to 2 mg/dl (less than or equal to 176.8 µmol/L)
* Adequate liver function, as evidenced by a serum bilirubin less than or equal to 1.5 times the laboratory normal range
* Hemoglobin greater than 11.0 g/dL
* Written informed consent (see Section 12.1)

Exclusion Criteria:

* Have had a Splenectomy for any reason
* Any known history of bone marrow stem cell disorder (Any abnormal bone marrow findings other than those typical of ITP must be approved by Amgen before a subject may be enrolled in the study)
* Any active malignancy. If prior history of cancer other than basal cell carcinoma or cervical carcinoma in situ, no treatment or active disease within 5 years before randomization
* Documented diagnosis of arterial thrombosis (i.e., stroke, transient ischemic attack or myocardial infarction) in the past year
* History of venous thrombosis (i.e., deep vein thrombosis, pulmonary embolism) including those subjects who are on ant-coagulation therapy
* Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure [NYHA greater than class II], uncontrolled hypertension [diastolic greater than 100 mmHg] or cardiac arrhythmia)
* Have 3 or more of the following predisposing factors for thromboembolic events: diabetes; smoker; using oral contraceptives; on estrogen therapy; known positive for anti-phospholipid antibodies; hypertriglyceridemia; hypercholesteremia (greater than 240 mg/dL); treatment for hypertension
* Known positive test for human immunodeficiency virus (HIV) infection or hepatitis C virus
* Currently receiving any treatment for ITP except corticosteroids, azathioprine or danazol administered at a constant dose and schedule
* IV Ig or anti-D Ig within 2 weeks before the screening visit
* Rituximab (for any indication) within 14 weeks before the screening visit or anticipated use during the time of the proposed study
* Received hematopoietic growth factors, including IL-11 (oprelvekin) within 4 weeks before the screening visit
* Past or present participation in any study evaluating PEG-rHuMGDF, recombinant human thrombopoietin (rHuTPO), AMG 531 or related platelet product
* Received any aklylating agents within 8 weeks before the screening visit or anticipated use during the time of the proposed study
* Less than 4 weeks since receipt of any therapeutic drug or device that is not FDA approved for any indication before the screening period - Less than 8 weeks since major surgery
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator
* Known hypersensitivity to any recombinant E coli-derived product
* Concerns for subject's compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-04-07 (Actual); Primary Completion 2006-12-01 (Actual); Study Completion 2007-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AMG 531 in the treatment of thrombocytopenia in subjects with ITP as measured by durable platelet response during the last 8 weeks of treatment and other platelet response parameters | Last 8 weeks of treatments

SECONDARY OUTCOMES:
To evaluate the overall safety of AMG 531 | Entire duration of the study including the follow up period
To evaluate possible reductions in the dose of concurrent ITP therapies while receiving AMG 531 | Entire duration of the study
To evaluate changes in Patient Reported Outcomes (PRO) and Health Resource Utilization (HRU) due to treatment with AMG 531 | Entire duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cines DB, Wasser J, Rodeghiero F, Chong BH, Steurer M, Provan D, Lyons R, Garcia-Chavez J, Carpenter N, Wang X, Eisen M. Safety and efficacy of romiplostim in splenectomized and nonsplenectomized patients with primary immune thrombocytopenia. Haematologica. 2017 Aug;102(8):1342-1351. doi: 10.3324/haematol.2016.161968. Epub 2017 Apr 14. PMID 28411254
- [Background] Kuter DJ, Newland A, Chong BH, Rodeghiero F, Romero MT, Pabinger I, Chen Y, Wang K, Mehta B, Eisen M. Romiplostim in adult patients with newly diagnosed or persistent immune thrombocytopenia (ITP) for up to 1 year and in those with chronic ITP for more than 1 year: a subgroup analysis of integrated data from completed romiplostim studies. Br J Haematol. 2019 May;185(3):503-513. doi: 10.1111/bjh.15803. Epub 2019 Feb 21. PMID 30793285
- [Background] Kuter DJ, Arnold DM, Rodeghiero F, Janssens A, Selleslag D, Bird R, Newland A, Mayer J, Wang K, Olie R. Safety and efficacy of self-administered romiplostim in patients with immune thrombocytopenia: Results of an integrated database of five clinical trials. Am J Hematol. 2020 Jun;95(6):643-651. doi: 10.1002/ajh.25776. Epub 2020 Mar 21. PMID 32129511
- [Derived] Weitz I, Sanz MA, Henry D, Schipperus M, Godeau B, Northridge K, Gleeson M, Danese M, Deuson R. A novel approach to the evaluation of bleeding-related episodes in patients with chronic immune thrombocytopenia. Curr Med Res Opin. 2012 May;28(5):789-96. doi: 10.1185/03007995.2012.684046. Epub 2012 Apr 25. PMID 22494019
- [Derived] Kuter DJ, Mufti GJ, Bain BJ, Hasserjian RP, Davis W, Rutstein M. Evaluation of bone marrow reticulin formation in chronic immune thrombocytopenia patients treated with romiplostim. Blood. 2009 Oct 29;114(18):3748-56. doi: 10.1182/blood-2009-05-224766. Epub 2009 Aug 11. PMID 19671919
- [Derived] Kuter DJ, Bussel JB, Lyons RM, Pullarkat V, Gernsheimer TB, Senecal FM, Aledort LM, George JN, Kessler CM, Sanz MA, Liebman HA, Slovick FT, de Wolf JT, Bourgeois E, Guthrie TH Jr, Newland A, Wasser JS, Hamburg SI, Grande C, Lefrere F, Lichtin AE, Tarantino MD, Terebelo HR, Viallard JF, Cuevas FJ, Go RS, Henry DH, Redner RL, Rice L, Schipperus MR, Guo DM, Nichol JL. Efficacy of romiplostim in patients with chronic immune thrombocytopenic purpura: a double-blind randomised controlled trial. Lancet. 2008 Feb 2;371(9610):395-403. doi: 10.1016/S0140-6736(08)60203-2. PMID 18242413
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_46_AMP-2_20030212.pdf
- See also: FDA-approved Drug Labeling — http://www.nplate.com/